CLINICAL TRIAL: NCT07192523
Title: Effect of Fluid Transfusion Regimens On Glycocalyx
Brief Title: Effects of Different Fluid Transfusion Regimens On Glycocalyx In Patients Undergoing Thoracic Surgery.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kocaeli Derince Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Tahsin Şimşek, ASSOCİATED PROFESSOR, Kocaeli Derince Education and Research Hospital
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: 2019/514/154/10
Record Dates: First submitted 2025-06-10; First posted 2025-09-25 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2026-01

CONDITIONS: Hypervolemia; Hypovolemia
Keywords: Endothelial Dysfunction
MeSH Terms: conditions — Edema; Hypovolemia | interventions — N-(2-aminophenyl)-6-(4-(2-(3,5-dihydroxycyclohexylidene)ethylidene)-7a-methyloctahydro-1H-inden-1-yl)-4-methylhepta-2,4-dienamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Effects of 3ml Fluid Transfusion Regimens On Glycocalyx (Other): In intraoperative fluid therapy, Group Restrictive received 3ml/kg/hr Ringer Lactate
  Interventions: Other: Restrictive fluid therapy
- Effects of 8 ml Fluid Transfusion Regimens On Glycocalyx (Other): In intraoperative fluid therapy, one group Group Liberal received 8ml/kg/hr crystalloid Ringer Lactate.
  Interventions: Other: Liberal fluid therapy

INTERVENTIONS:
Other: Restrictive fluid therapy — Group Restrictive (Group R) received 3ml/kg/hr, crystalloid (Ringer Lactate).
  Other Names: 3 ml
  Arms: Effects of 3ml Fluid Transfusion Regimens On Glycocalyx
Other: Liberal fluid therapy — Group Restrictive liberal received 8ml/kg/hr, crystalloid (Ringer Lactate).
  Other Names: 8 ml
  Arms: Effects of 8 ml Fluid Transfusion Regimens On Glycocalyx

SUMMARY:
Introduction: Endothelial Glycocalyx (EG) composing of proteoglycans heparan sulfate (HS), syndecan, and plasma proteins forms a physiologically active surface layer on the vascular endothelium, regulates oncotic pressure. We aimed to compare the effects of two different fluid transfusion regimens on EG.

Materials and Methods: 41 patients with ASA I-III physical status were included in this prospective, randomized controlled study. We collected blood samples before anesthesia induction and after surgery to measure hemoglobin-hematocrit levels and biochemical parameters. Hemodynamic parameters were recorded every 15 minutes perioperatively. We divided the patients into two groups: Group R received 3 ml/kg/h, and Group L received 8 ml/kg/h of Ringer's lactate infusion. To assess endothelial damage, HS and syndecan levels, blood samples were taken after anesthesia induction(T1), after pneumonectomy or lobectomy(T2), and at the end of surgery(T3).

DETAILED DESCRIPTION:
This prospective, randomized-controlled study was conducted between August 15, 2021, and December 15, 2021, at a University Hospital. Local ethics committee approval (protocol no: 2019/514/154/10) was obtained for the study. The study was conducted in accordance with the Declaration of Helsinki. Written and verbal consent was obtained from all patients included in the study.

Participants 41 patients who underwent elective thoracic surgery were included in the study. Inclusion criteria; being 18-65 years old and in the American Society of Anaesthesiologists (ASA) I-III risk group. Exclusion criteria from the study were determined as not accepting to participate in the study, having heart failure, having a previously known vascular disease, and having more than 500 ml of blood replacement during the perioperative period.

Anesthesia protocol Patients were restricted from consuming solid and semi-solid food 6 hours before the operation. Water consumption was allowed until 2 hours before the operation. After all patients were taken to the operation room, standard monitoring techniques including electrocardiogram (ECG), pulse oximetry (SpO2), end-tidal carbon dioxide pressure (ETCO2), non-invasive blood pressure and body temperature monitoring were applied, and a Foley urinary catheter was inserted. After a 25 G intravenous (iv) catheter was opened on the back of the hand, 1-1.5 mg/kg propofol, 1-2 mcg/kg fentanyl and 0.6 mg/kg rocuronium were administered for general anesthesia induction, and tracheal intubation was performed with a No. 7.5 double lumen tracheal tube. After intubation, fresh gas flow was adjusted to 2lt/min (50% oxygen and 50% air). For maintenance of anesthesia, sevoflurane was titrated at a concentration of 2-2.5% to maintain MAC 1 and BIS 40-60. In intraoperative fluid therapy, one group (Group Restrictive (Group R)) received 3ml/kg/hr, and the other group (Group Liberal (Group L)) received 8ml/kg/hr crystalloid (Ringer Lactate). Blood replacement was applied according to the hemodynamic data and bleeding amounts of the patients. Blood samples were taken from the patients for hemogram, BUN, and creatinine measurements before and after surgery. Twenty minutes before the end of the operation, all patients were administered tramadol 100 mg and paracetamol 1 gr intravenously for postoperative analgesia. After the end of the surgery, 0.015 mg/kg atropine and 0.04 mg/kg neostigmine were administered to the patients for decurarization. Following extubation with adequate muscle strength and spontaneous ventilation, the patients were taken to the postoperative care unit.

Collection of Blood Samples To evaluate endothelial damage, blood samples were taken from patients in both groups 3 times. The time of taking the samples was determined as; the blood sample taken after the placement of the IV cannula (T1), the blood sample taken after pneumonectomy or lobectomy (T2), and the blood sample taken after the patient was extubated following the end of surgery (T3). Venous blood samples were placed in a 5 ml vacuum tube with a serum separator. The samples were centrifuged at 1500 g for 10 minutes to separate the serum, and these samples were stored at -80 °C.

Biochemical analysis Studies for the analysis of heparan sulfate and syndecan phosphate parameters were carried out in the Medical Biochemistry Laboratory of our University Faculty of Medicine. The serum concentration of Syndecan-1 was determined using the enzyme-linked immunosorbent assay (ELISA) technique. Serum syndecan-1 levels were analyzed using an ELISA kit (catalog no. E3344Hu.), purchased from BT-laboratory. Ltd. (City, China) following the manufacturer's instructions, and the results are expressed in ng/ml. The intra-assay coefficient of variation (CV) of Syndecan-1 was <8% and the inter-assay CV was <10% for this parameter.

ELIGIBILITY:
Inclusion Criteria:

. Being 18-65 years old and in the American Society of Anaesthesiologists (ASA) I-III risk group.

Exclusion Criteria:

* Having heart failure
* Having a previously known vascular disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2021-08-15 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2025-08-30 (Actual)

PRIMARY OUTCOMES:
Our primary aim in the study was to evaluate the changes in HS and syndecan 1 levels after 8 ml/kg/hr or 3 ml/kg/hr fluid transfusion in thoracic surgery. | 6 month
  To evaluate endothelial damage, blood samples were taken from patients in both groups 3 times. The time of taking the samples was determined as; the blood sample taken after the placement of the IV cannula (T1), the blood sample taken after pneumonectomy or lobectomy (T2), and the blood sample taken after the patient was extubated following the end of surgery (T3). Venous blood samples were placed in a 5 ml vacuum tube with a serum separator. The samples were centrifuged at 1500 g for 10 minutes to separate the serum, and these samples were stored at -80 °C.

CONTACTS AND LOCATIONS:
Locations (1):
- Kartal Dr Lutfi Kirdar City Hospital, Istanbul, Kartal, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No